CLINICAL TRIAL: NCT06303219
Title: Comparative Effects of Traditional Moderate Intensity Training and High Intensity Interval Training on Anxiety, Fatigue and Quality of Life in Polycystic Ovarian Syndrome
Brief Title: Effects of Traditional Moderate Intensity Training and High Intensity Interval Training in Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0577
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: Anxiety; Fatigue; High Intensity Interval Training; Polycystic Ovarian Syndrome; Quality of Life.
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anxiety Disorders; Fatigue | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRADITIONAL MODERATE INTENSITY TRAINING (Experimental)
  Interventions: Other: RADITIONAL MODERATE INTENSITY TRAINING
- HIGH INTENSITY INTERVAL TRAINING (Active Comparator)
  Interventions: Other: HIGH INTENSITY INTERVAL TRAINING

INTERVENTIONS:
Other: RADITIONAL MODERATE INTENSITY TRAINING — It consists of patients who will receive High-intensity interval training, including running as well as walking at 80% to 95% HR peak. Which is monitored by a smart watch. Before starting treatment, it follows a 10-minute warm-up exercise which includes basic stretches (Quads, Hams, and calf muscles) with a 30-second hold of both legs and same exercise will be pursued for the cool-down period. This intervention will be performed 5 days per week for 4 weeks.
  The total duration of this session will be 50 minutes
  Arms: TRADITIONAL MODERATE INTENSITY TRAINING
Other: HIGH INTENSITY INTERVAL TRAINING — It consists of patients who will receive Moderate-intensity interval training, including running as well as walking at 60% HR peak. Which is monitored by a smart watch. Before starting treatment, it follows a 10-minute warm-up exercise which includes basic stretches (Quads, Hams, and calf muscles) with a 30-second hold of both legs and same exercise will be pursued for the cool-down period. This intervention will be performed 5 days per week for 4 weeks.
  The total duration of this session will be 50 minutes (
  Arms: HIGH INTENSITY INTERVAL TRAINING

SUMMARY:
To determine the comparative effects of traditional moderate intensity training and high intensity interval training on Anxiety, fatigue and Quality of Life in females with polycystic ovarian syndrome

ELIGIBILITY:
Inclusion Criteria:

* Participants with BMI greater than 25kg/m2
* Oligo- or anovulation/irregular cycles i.e 35 days
* Married women
* Primary infertility
* A diagnosis of polycystic ovaries based on ultrasound results

Exclusion Criteria:

* Use of psychiatric or psychotropic medications.
* Unresolved gynecological conditions i.e Cervical Dysplasia, Pelvic floor prolapse, Uterine Fibroids, Urinary Incontinence
* Diabetes, pregnancy, smoking, illness or injury that prevented or limited exercise performance and existing participation in regular physical activity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POLYCYSTIC OVARIAN SYNDROME
Enrollment: 44 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating scale (HAM-A) | 4th week
  The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms, and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Although the HAM-A remains widely used as an outcome measure in clinical trials. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Reliability and concurrent validity of the HAM-A and its subscales were sufficient. The Cronbach's α of the Hamilton Anxiety Scale was 0.89
The Polycystic Ovary Syndrome Health-Related Quality of Life Questionnaire (PCOSQ) | 4th week
  The PCOSQ consists of five domains, each relating to a common symptom of PCOS; body hair, emotions, infertility, menstrual problems and infertility. Each question on the PCOSQ is associated with a 7-point scale in which 7 represents optimal function and 1 the poorest function. All five PCOSQ dimensions were internally reliable with Cronbach's alpha scores ranging from 0.70 to 0.97. Intra-class correlation coefficients to evaluate test-retest reliability were high (range 0.89-0.95, P < 0.001). All five PCOSQ dimensions were internally reliable with Cronbach's α scores ranging from 0.70 to 0.97. Construct validity was demonstrated by high correlations for PCOSQ (0.49 and 0.54)
The Fatigue Impact Scale (FIS) | 4th week
  The FIS was developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. Daily Fatigue Impact Scale (D-FIS) consist of eight items that could be used for monitoring daily changes in fatigue. The test-retest reliability of FIS was good in terms of its cognitive, physical, and psychosocial subscales and total scores, with ICC values of 0.78, 0.73, 0.80, and 0.83, respectively

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, Principal Investigator — Riphah International University
Locations (1):
- Gynecological Department of Fatima Memorial Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kite C, Lahart IM, Afzal I, Broom DR, Randeva H, Kyrou I, Brown JE. Exercise, or exercise and diet for the management of polycystic ovary syndrome: a systematic review and meta-analysis. Syst Rev. 2019 Feb 12;8(1):51. doi: 10.1186/s13643-019-0962-3. PMID 30755271
- [Background] Teede HJ, Tay CT, Laven JJE, Dokras A, Moran LJ, Piltonen TT, Costello MF, Boivin J, Redman LM, Boyle JA, Norman RJ, Mousa A, Joham AE; International PCOS Network. Recommendations from the 2023 international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Eur J Endocrinol. 2023 Aug 2;189(2):G43-G64. doi: 10.1093/ejendo/lvad096. PMID 37580861
- [Background] Patten RK, Bourke M, McIlvenna LC, Moreno-Asso A, Woessner MN, Stepto NK, Parker A. Longitudinal affective response to high-intensity interval training and moderate-intensity continuous training in overweight women with polycystic ovary syndrome: A randomised trial. Psychol Sport Exerc. 2023 Jan;64:102325. doi: 10.1016/j.psychsport.2022.102325. Epub 2022 Oct 26. PMID 37665810
- [Background] Patten RK, McIlvenna LC, Levinger I, Garnham AP, Shorakae S, Parker AG, McAinch AJ, Rodgers RJ, Hiam D, Moreno-Asso A, Stepto NK. High-intensity training elicits greater improvements in cardio-metabolic and reproductive outcomes than moderate-intensity training in women with polycystic ovary syndrome: a randomized clinical trial. Hum Reprod. 2022 May 3;37(5):1018-1029. doi: 10.1093/humrep/deac047. PMID 35325125
- [Background] Kite C, Parkes E, Taylor SR, Davies RW, Lagojda L, Brown JE, Broom DR, Kyrou I, Randeva HS. Time to Load Up-Resistance Training Can Improve the Health of Women with Polycystic Ovary Syndrome (PCOS): A Scoping Review. Med Sci (Basel). 2022 Sep 22;10(4):53. doi: 10.3390/medsci10040053. PMID 36278523
- [Background] Patel V, Menezes H, Menezes C, Bouwer S, Bostick-Smith CA, Speelman DL. Regular Mindful Yoga Practice as a Method to Improve Androgen Levels in Women With Polycystic Ovary Syndrome: A Randomized, Controlled Trial. J Am Osteopath Assoc. 2020 Apr 14. doi: 10.7556/jaoa.2020.050. Online ahead of print. PMID 32285088
- [Background] Abdollahi L, Mirghafourvand M, Babapour JK, Mohammadi M. Effectiveness of cognitive-behavioral therapy (CBT) in improving the quality of life and psychological fatigue in women with polycystic ovarian syndrome: a randomized controlled clinical trial. J Psychosom Obstet Gynaecol. 2019 Dec;40(4):283-293. doi: 10.1080/0167482X.2018.1502265. Epub 2018 Sep 3. PMID 30175648
- [Background] .Jakhar R, Sen ED, Rastogi P. Improvement In Health-Related Quality of Life in Polycystic Ovarian Syndrome: A Randomized Controlled Trial. Journal of Survey in Fisheries Sciences. 2023:382-8.
- [Background] Ashila A, Murugaraj T. Effect of High Intensity Interval Training on Body Mass Index, Plasma Glucose and Insulin Among Individuals with Polycystic Ovary Syndrome Living in the South Indian Coast. Journal of Coastal Life Medicine. 2023;11:2579-85